CLINICAL TRIAL: NCT05130255
Title: Phase 1 Trial With GD2-SADA:177Lu-DOTA Drug Complex in Patients With Recurrent or Refractory Metastatic Solid Tumors Known to Express GD2, Including Small Cell Lung Cancer, High Risk Neuroblastoma, Sarcoma and Malignant Melanoma
Brief Title: GD2-SADA:177Lu-DOTA Complex in Patients With Solid Tumors Known to Express GD2
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1001
Record Dates: First submitted 2021-11-11; First posted 2021-11-23 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: SCLC; Malignant Melanoma; Sarcoma; High Risk Neuroblastoma
MeSH Terms: conditions — Melanoma; Sarcoma

STUDY DESIGN:
Intervention Model Description: Phase 1 dose-escalation single-arm, open-label, non-randomized, multi-center trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GD2-SADA:177Lu-DOTA Complex (Experimental): GD2-SADA IV. infusion followed by 177Lu-DOTA IV. infusion (The IMP is a two-step radioimmunotherapy, delivered as two separate products GD2-SADA and 177Lu-DOTA ).
  1 treatment cycle in Part A, 2 treatment cycles in Part B and up to 5 treatment cycles in Part C
  Interventions: Drug: GD2-SADA:177Lu-DOTA Complex

INTERVENTIONS:
Drug: GD2-SADA:177Lu-DOTA Complex — The IMP is a two-step radioimmunotherapy, delivered as two separate products GD2-SADA and 177Lu-DOTA, both will be administered as an IV infusion
  Other Names: two-step radioimmunotherapy

SUMMARY:
Patients with Small Cell Lung Cancer, High Risk Neuroblastoma, Sarcoma and Malignant Melanoma will be treated with GD2-SADA:177Lu-DOTA complex(The IMP is a two-step radioimmunotherapy, delivered as two separate products GD2-SADA and 177Lu-DOTA) to assess safety and tolerability

DETAILED DESCRIPTION:
A phase 1 dose-escalation single-arm, open-label, non-randomized, multi-center trial of the safety and tolerability of GD2-SADA:177Lu-DOTA complex in GD2 expressing solid tumors.

The trial is planned as a Phase 1 trial with three parts, A, B and C. Escalation in this trial will be based on a classical 3+3 trial design.

Part A is a GD2-SADA dose escalation phase, in which patients will receive one treatment cycle.

Part B is a 177Lu-DOTA dose escalation phase, in which patients will receive up to 2 treatment cycles .

Part C is a repeated dosing phase where the doses determined in Part A and B will be administered. Patients will receive repeated treatment cycles with a maximum of 5 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from patient, legal guardian(s) and/or adolescents obtained in accordance with local regulations. Pediatric patients must provide assent as required by local regulations.
* Age ≥18 years at the time of informed consent, for High Risk Neuroblastoma & sarcoma age ≥16 years of age at time of informed consent/assent
* Measurable disease according to RECIST 1.1
* ECOG performance status 0-1
* Expected survival >3 months
* Platelet counts ≥100,000 cells/mm3
* Hemoglobin ≥9 g/dL
* Adequate renal function with serum creatinine ≤1.5 mg/dL or creatinine clearance ≥60mL/min as calculated using the Cockcroft-Gault equation
* Patient willing and able to comply with the trial protocol

Exclusion Criteria:

* Systemic chemotherapy, radiotherapy, immunotherapy, or major surgery administered within 3 weeks prior to the first planned dosing of the IMP per protocol
* Patients receiving any other investigational therapy for their cancer within 3 weeks prior to the first planned dosing of the IMP per protocol
* Ongoing radiation toxicities from prior RT therapy
* Patients with a diagnosis of autoimmune diseases or immunodeficiencies or documented infection with human immunodeficiency virus (HIV) or hepatitis B or C virus (active)
* Prior treatment with anti-GD2 antibody

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
To determine the optimal, safe GD2-SADA protein dose and dosing interval between GD2-SADA and 177Lu-DOTA administrations | 6 weeks
  Occurrence of DLTs (Part A)
To determine maximum tolerable activity of 177Lu-DOTA | 6 weeks
  Occurrence of DLTs (Part B)
To assess cumulative toxicity signals and safety profile (Number and severity of adverse events) following repeated dosing and determine the recommended phase 2 dose (RP2D) | 52 weeks
  Number and severity of adverse events (Part C)

CONTACTS AND LOCATIONS:
Overall Officials: Taofeek K Owonikoko, MD/PhD, Principal Investigator — University of Maryland, Marlene & Steward Greenebaum Comprehensive Cancer Center 22 S Greene St, Baltimore, MD 21201
Locations (8):
- United States (8):
  - HonorHealth, Scottsdale, Arizona
  - City of Hope National Medical Center, Duarte, California
  - University of Chicago, Chicago, Illinois
  - Corewell Health-BAMF Health, Grand Rapids, Michigan
  - Memorial Sloan- Kettering Cancer Center, New York, New York
  - Case Western Reserve University, Cleveland, Cleveland, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided